CLINICAL TRIAL: NCT06491381
Title: Incidence of Post Cesarean Section Wound Infections At Emergency Unit At E-Hhussien University Hospital
Brief Title: Post Cesarian Section Wound Infections At Emergency Room
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Muhamed Ahmed Abdelmoaty Muhamed Alhagrasy, Dr., Al-Azhar University
Other Study IDs: obstet1724
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Surgical Wound Infection
Keywords: Surgical site infections; Elective Cesarean delivery; Emergency Room
MeSH Terms: conditions — Surgical Wound Infection; Emergencies | interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Elective Cesarean Delivery: This group will consist of 110 patients who are scheduled for planned cesarean deliveries at El-hussien Hospital. These patients will have non-emergency indications for cesarean section, such as previous cesarean delivery, breech presentation, maternal request, or other medical indications that allow for scheduled surgery. Participants in this group will undergo standard pre-operative preparation and receive routine post-operative care as per hospital protocols. Their surgical site will be monitored for signs of infection during their hospital stay and follow-up period.
  Interventions: Procedure: Cesarean delivery
- Emergency Cesarean Delivery: This group will consist of 110 patients who undergo unplanned, emergency cesarean deliveries at the Emergency Unit of El-hussien Hospital. Indications for emergency cesarean section may include, but are not limited to, fetal distress, placental abruption, cord prolapse, failed induction of labor, or arrest of labor progression. Patients with premature rupture of membranes will be excluded from this group due to their increased risk of infection. Participants in this group will receive urgent pre-operative preparation and post-operative care as per hospital emergency protocols. Their surgical sites will be monitored for signs of infection during their hospital stay and follow-up period, similar to the elective group.
  Interventions: Procedure: Cesarean delivery

INTERVENTIONS:
Procedure: Cesarean delivery — The cesarean section will begin with a Pfannenstiel incision above the pubic bone, followed by blunt dissection to separate tissue layers and retracting the rectus muscles for peritoneal cavity access. A transverse or vertical peritoneal incision will expose the uterus, and a transverse incision on the lower uterine segment will be made for delivery. The baby will be delivered, the umbilical cord clamped and cut, and the baby handed to the pediatric team. The placenta will be detached and delivered, and the uterus will be closed with multiple layers of sutures. The abdominal layers will be closed with absorbable Polyglactin (Vicryl) sutures for the rectus sheath and subcutaneous tissue, and non-absorbable Polypropylene sutures for the skin. A sterile dressing will be applied to protect the wound and promote a clean healing environment, ensuring proper surgical technique, tissue handling, and minimizing post-operative complications.

SUMMARY:
The goal of this observational study is to compare the incidence of post-cesarean section wound infections between emergency and elective cesarean deliveries at El-hussien Hospital. The main questions it aims to answer are:

Is there a difference in surgical site infection rates between emergency and elective cesarean sections? What are the other outcome measures associated with emergency versus elective cesarean deliveries?

Participants will be 220 patients undergoing cesarean section, divided into two groups:

110 patients undergoing emergency cesarean delivery in the Emergency Unit 110 patients undergoing elective cesarean delivery

Researchers will compare the emergency cesarean group to the elective cesarean group to see if there are differences in surgical site infection rates and other relevant outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Managed with elective CS or Emergency CS
* BMI < 25 Kg/m2

Exclusion Criteria:

* Immunodeficiency or diabetes.
* Premature rupture of membrane
* Bleeding disorder.
* Previous uterine surgery except previous CS.
* Malignancy.
* Refusal to participate.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study is open to female participants only. The inclusion of only female participants is due to the nature of the study, which focuses on cesarean section deliveries. Cesarean sections are surgical procedures performed exclusively on pregnant women to deliver their babies. As pregnancy and childbirth are biological processes unique to individuals with female reproductive organs, male participants are not eligible for this study.
Study Population: This study will include 220 patients undergoing cesarean section at El-hussien Hospital, equally divided into two groups of 110 each. One group will consist of emergency cesarean deliveries performed in the Emergency Unit, excluding cases with premature rupture of membranes. The other group will include elective, scheduled cesarean deliveries. This diverse population will allow for a comprehensive comparison of surgical site infection rates and other outcomes between emergency and elective cesarean sections.
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Post Caesarian Section Wound Infections | 6 weeks after surgery.
  * The wounds will be inspected. The presence of minor or major wound infection will be recorded on an audit form.
  * Wound infection will be defined as:
  Purulent discharge present within or exuding from the wound. Painful spreading erythema indicative of cellulitis.
  • An infection will be defined as minor if deep tissue destruction or lymphangitis is absent, and major if these elements, wound dehiscence or systemic symptoms, is present.

SECONDARY OUTCOMES:
Wound Healing Complications | 6 weeks after surgery.
  We will assess the occurrence of other wound-related complications, such as wound dehiscence (separation of wound edges), seroma (accumulation of fluid), or hematoma (collection of blood).
Length of Hospital Stay | 6 weeks after surgery.
  We will measure the duration of hospitalization for patients who undergo a cesarean section at the emergency unit and hospital.
Surgical Site Pain | 6 weeks after surgery.
  We will evaluate the intensity and duration of pain experienced by patients at the surgical site following a cesarean section.
Antibiotic Usage | 6 weeks after surgery.
  We will measure the frequency, type, and duration of antibiotic administration to treat post-cesarean section wound infections.
Patient Satisfaction | 6 weeks after surgery.
  We will assess the level of satisfaction reported by patients regarding their overall experience with the cesarean section procedure and subsequent wound healing.
Keloid formation | 6 months after the surgery
  We will assess formation of keloid after the surgery/

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Hussein University Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified individual participant data (IPD) from this study. The shared data will include baseline demographics, clinical characteristics, surgical details, and outcome measures related to surgical site infections and other relevant outcomes for both emergency and elective cesarean section groups.
  Data will be available beginning 9 months after the main study results are published. Researchers who provide a methodologically sound proposal will be allowed access to the data. Proposals should be directed to the corresponding author. The corresponding author will also be responsible for making the data available to approved researchers.
  To gain access, data requestors will need to sign a data access agreement. The data will be available for 5 years for researchers whose proposed use of the data has been approved. The shared dataset will exclude participant identifying information and comply with privacy regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available beginning 9 months after the main study results are published. Researchers who provide a methodologically sound proposal will be allowed access to the data. Proposals should be directed to the corresponding author. The corresponding author will also be responsible for making the data available to approved researchers.
  To gain access, data requestors will need to sign a data access agreement. The data will be available for 5 years for researchers whose proposed use of the data has been approved.
Access Criteria: Researchers must submit a written proposal to the corresponding author outlining the research questions, methodology, team qualifications, and potential impact. Proposals will be reviewed based on scientific merit, compatibility with original study objectives, feasibility, and potential to advance medical knowledge or patient care. Requestors must agree to use the data only for the approved purpose, maintain confidentiality and security, not identify or contact participants, and acknowledge the original study in publications. Researchers must sign a data use agreement covering data access terms, security, publication guidelines, and result sharing with the original team. Priority may be given to early career researchers, those from low- and middle-income countries, and collaborative projects. The corresponding author reserves the right to deny access if criteria are not met or if there are concerns about responsible data use.